CLINICAL TRIAL: NCT06121531
Title: A Prospective, Randomized, Double-blind, Parallel, Active-controlled Clinical Study of Silicone Hydrogel Monthly Soft Contact Lens for the Safety and Effectiveness in Visual Correction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yung Sheng Optical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0438TC01
Record Dates: First submitted 2023-10-30; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Contact Lenses, Hydrophilic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Active Comparator): Si-Hy (Samfilcon A)
  Interventions: Device: Soft Contact Lens
- Group II (Experimental): Si-Hy (Otufilcon A)
  Interventions: Device: Soft Contact Lens

INTERVENTIONS:
Device: Soft Contact Lens — Vision Correction

SUMMARY:
This was a prospective, randomized, double-blind, parallel, active-controlled clinical study to assess the safety and efficacy of Silicone Hydrogel Contact Lens for vision correction.

ELIGIBILITY:
Inclusion Criteria:

1. 20 years old and above.
2. Subjects with normal eyes who are not using any ocular medications (excluding ocular lubricants and artificial tears).
3. Best spectacle corrected visual acuity greater than or equal to 1.0 for both eyes.
4. With +6.00D ~ -12.00 D spherical power, and ≦1.00 D astigmatism (based on subjective optometry measurements).
5. Have worn soft contact lens for at least 1 month prior to the study.
6. Willing to comply with the required wearing time and use specified contact lens care product.
7. Agree to comply with all study procedures and signed the informed consent form before enrollment.

Exclusion Criteria:

1. Anterior chamber infection, inflammation, or abnormality.
2. Any active ocular disease that would affect contact lens wear or vision (such as acute and subacute inflammation of the anterior chamber of the eye, eye infection, uveitis, serious palpebral abnormality, corneal hypoesthesia, corneal epithelium abrasion, dry eye and tear duct defection, ocular allergies, highly suspected glaucoma) upon evaluation by the investigators or slit lamp findings.
3. Currently using systemic or ocular medications that would contraindicate with contact lens wear (such as, glaucoma eye drops, steroid anti-inflammatory drops, eye ointments, eye gels and other eye medicines).
4. History of herpes simplex keratitis.
5. History of refractive surgery, keratoconus, or irregular cornea.
6. Slit lamp findings that are not suitable for inclusion (Details of the grading standards for each eye condition are specified in CIP section 5.7.5 from page 38 to 43).
7. A pathologically dry eye syndrome (Schirmer test < 5 mm).
8. Have participated in any contact lens or contact lens care product clinical trials within the previous 1 month (excluding questionnaire types and specimen collection).
9. Currently pregnant or lactation.
10. Allergy to any contact lens care product ingredient (such as mercury or topical antimicrobial agent).
11. Have experienced discomfort when wearing hydrogel contact lens.
12. Subjects who are judged unsuitable for the study by the investigators.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 144 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
The effectiveness of corrected visual acuity | 3 Months
  The effectiveness of corrected visual acuity at 3-month. Effectiveness is defined as visual acuities of both eyes correctable to ≥1.0 with contact lens.
  Effectiveness formula (%): total number of subjects with vision correction of ≥ 1.0 at a given timepoint / total number of subjects enrolled at a given time × 100 %.
  Definition of total number of subjects enrolled at a given time: the total number of subjects conforming to the PPS criteria and having worn lenses for 3 months.

SECONDARY OUTCOMES:
Effectiveness of corrected visual acuity | 1 week, 1 month and 2 months
  Effectiveness of corrected visual acuity at 1 week, 1 month and 2 months. The effectiveness (%) is defined as total number of subjects with vision correction of ≥ 1.0 at a given timepoint / total number of subjects enrolled at a given time × 100 %.
Average contact lens corrected visual acuity | 1 week, 1 month, 2 months and 3 months
  The mean, standard deviation, median, maximum, minimum, Q1, Q3 and Inter-Quartile Range (IQR) will be calculated for "Lens corrected visual acuity". Comparisons between the Treatment group and Control group will be made.
Change in diopter (Spherical and cylindrical power of subjective optometry) | 1 week, 1 month, 2 months and 3 months
  The mean, standard deviation, median, maximum, minimum, Q1, Q3 and Inter-Quartile Range (IQR) will be calculated for "power" (the spherical and cylindrical power). Comparisons between the Treatment group and Control group will be made.
Change in corneal astigmatism (the vertical and horizontal keratometry meridian, the power and axis of astigmatism) | 1 week, 1 month, 2 months and 3 months
  The mean, standard deviation, median, maximum, minimum, Q1, Q3, and Inter-Quartile Range (IQR) will be calculated for "corneal astigmatism" (the vertical and horizontal curvature, the power and axis of astigmatism).
  Comparisons between the Treatment group and Control group will be made.
Lens broken rate | 1 week, 1 month, 2 months and 3 months
  The number and percentage of parameters (total lenses, unbroken lenses, broken lenses) will be calculated and analyzed.
  Comparisons between the Treatment group and Control group will be made.
Lens fitting (lens centration, lens movement, coverage, and tightness) | 1 week, 1 month, 2 months and 3 months
  The total number and percentage of parameters (lens centration, lens movement, coverage, tightness) with grading scale evaluated by investigators will be calculated and analyzed.
  Comparisons between the Treatment group and Control group will be made.
Subjective acceptance (comfort, vision, lens handling, lens cleaning) | 1 week, 1 month, 2 months and 3 months
  The total number and percentage of parameters (comfort, vision, lens handling, lens cleaning) with a grading scale using questionnaires will be calculated and analyzed.
  Comparisons between the Treatment group and Control group will be made.
Lens state (lens front surface wettability, front surface deposits, back surface deposits) | 1 week, 1 month, 2 months and 3 months
  The total number and percentage of parameters (lens front surface wettability, front surface deposits, back surface deposits) with a grading scale evaluated by investigators will be calculated and analyzed.
  Comparisons between the Treatment group and Control group will be made.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Tri-Service General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District